CLINICAL TRIAL: NCT07325903
Title: Research of Integrated Traditional Chinese and Western Medicine on Precocious Puberty
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDCH-ZY-2025402
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Puberty, Precocious
Keywords: precocious puberty; Sanghe Jianghuo Granules; RCT
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 10% drug-containing placebo, for a period of 3 months.
  Interventions: Combination Product: 10% drug-containing placebo, for a period of 3 months.
- Intervention group (Active Comparator): administered "Mulberry and Lotus Leaf Heat-Clearing Granules," with the following drug composition: mulberry leaves, lotus leaves, fresh rehmannia, anemarrhena, scutellaria, atractylodes, etc., for an intervention period of 3 months..
  Interventions: Drug: administered "Mulberry and Lotus Leaf Heat-Clearing Granules," with the following drug composition: mulberry leaves, lotus leaves, fresh rehmannia, anemarrhena, scutellaria, atractylodes, etc.

INTERVENTIONS:
Drug: administered "Mulberry and Lotus Leaf Heat-Clearing Granules," with the following drug composition: mulberry leaves, lotus leaves, fresh rehmannia, anemarrhena, scutellaria, atractylodes, etc. — administered "Mulberry and Lotus Leaf Heat-Clearing Granules," with the following drug composition: mulberry leaves, lotus leaves, fresh rehmannia, anemarrhena, scutellaria, atractylodes, etc., for an intervention period of 3 months.
  Arms: Intervention group
Combination Product: 10% drug-containing placebo, for a period of 3 months. — 10% drug-containing placebo, for a period of 3 months. The drug was Mulberry and Lotus Leaf Heat-Clearing Granules.
  Arms: Control group

SUMMARY:
Precocious puberty is characterized by the premature appearance of secondary sexual characteristics. Globally, the timing of puberty onset in children has shown a certain tendency to advance. In China, the incidence of precocious puberty has been increasing year by year. Precocious puberty exerts long-term and systemic impacts on children's health: advanced bone age leads to short stature; earlier sexual development than peers may induce emotional problems such as anxiety and inferiority; it may increase the risk of obesity and type 2 diabetes, posing long-term hazards to cardiovascular health; it may also result in irregular menstruation or dysmenorrhea, exerting indirect effects on reproductive health.

Modern traditional Chinese medicine (TCM) holds that: various factors lead to liver-kidney yin deficiency, hyperactivity of ministerial fire, and early arrival of tian gui (the substance responsible for promoting growth, development and reproduction), thereby triggering premature sexual development. The main syndrome types identified in clinical practice include yin deficiency with fire hyperactivity syndrome, liver stagnation transforming into fire syndrome, and phlegm-dampness internal accumulation syndrome.

Since the late 1970s, the investigators' department has taken the lead in treating precocious puberty with TCM diagnostic methods, proposing that the pathogenesis of precocious puberty lies in "kidney yin deficiency and hyperactivity of ministerial fire", and adopting the therapy of nourishing yin and purging fire for its treatment. A number of studies have confirmed that TCM medicines with the effects of nourishing yin and purging fire can effectively alleviate the yin deficiency with fire hyperactivity syndrome in children, delay the development of secondary sexual characteristics and bone age.

At present, central precocious puberty is mostly treated with gonadotropin-releasing hormone analogs (GnRHa). However, this treatment has the drawback of inhibiting the growth axis, yielding limited benefits for children with advanced bone age, overweight or obesity, and may even affect glucose and lipid metabolism. Moreover, some children with precocious puberty complicated with obesity may be intolerant to this therapy. In contrast, TCM therapy and integrated TCM-Western medicine therapy can effectively delay the development of secondary sexual characteristics and advanced bone age, and improve final adult height, thus being widely applied in China.

Although a large number of relevant studies have been reported in recent years and TCM diagnosis and treatment guidelines for precocious puberty have been formulated, there is still a lack of high-quality evidence-based medical research to support the advantageous aspects of integrated TCM-Western medicine diagnosis and treatment. Additionally, the underlying mechanisms of diagnosis and treatment for different syndrome types of precocious puberty remain insufficiently studied.

In this study, the investigators will conduct a multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the effects of Sanghe Jianghuo Granules on the regulation of the hypothalamic-pituitary-gonadal (HPG) axis, metabolic homeostasis and inflammatory microenvironment, so as to verify its efficacy and safety. Furthermore, combined with transcriptomics, proteomics and network pharmacology, the investigators will identify the key targets and action pathways of Sanghe Jianghuo Granules, and verify its regulatory effect on the HPG axis through in vivo and in vitro experiments.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients clinically diagnosed with precocious puberty: girls who exhibit secondary sexual characteristics or gonadal development before the age of 8, accompanied by obesity (BMI ≥ P85), and classified as having a syndrome of yin deficiency with hyperactivity of fire complicated by phlegm-dampness. Inclusion age: girls aged 5 years to 9 years, all of whom are initial cases and have not received any drug treatment related to precocious puberty.

Exclusion Criteria:

* Secondary precocious puberty, associated with diabetes, thyroid dysfunction, other endocrine disorders, and severe underlying conditions.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast Tanner Stages | The measurement times are before the start of the experiment and the 3rd month after the start
  Measured by the attending physician

SECONDARY OUTCOMES:
Bone age | The measurement times are before the start of the experiment and the 3rd month after the start
  Bone age is determined by radiologists in our hospital who take a posteroanterior radiograph of the left hand and judge the bone age according to the Greulich-Pyle (GP) atlas method.
Traditional Chinese Medicine syndrome score | The measurement times are before the start of the experiment and the 3rd month after the start
  Based on the Guidelines for Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment of Pediatric Precocious Puberty (2023 Edition) and clinical experience, the Traditional Chinese Medicine (TCM) syndrome scores were screened and determined.

OTHER OUTCOMES:
Testosterone | The measurement times are before the start of the experiment and the 3rd month after the start
  Testosterone(nmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
PRL | The measurement times are before the start of the experiment and the 3rd month after the start
  Prolactin(mIU/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Estradiol | The measurement times are before the start of the experiment and the 3rd month after the start
  Estradiol(pmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
FSH | The measurement times are before the start of the experiment and the 3rd month after the start
  Follicle-Stimulating Hormone(U/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
LH | The measurement times are before the start of the experiment and the 3rd month after the start
  Luteinizing Hormone(U/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Height | The measurement times are before the start of the experiment and the 3rd month after the start
  The height is measured and obtained by the physician. Place the mechanical height measuring device horizontally on a flat surface, against a wall, and calibrate the height measuring device reading. Instruct the examinee to stand barefoot on the base plate of the height measuring device, facing away from the pillar. When the doctor moves the height measuring device, he holds the handle of the height measuring device, moves horizontally, tries to keep the head upright, and keeps the body and limbs naturally straight. For hair knots and braids that are not convenient to measure height, they should be untied and headwear should be removed. The horizontal pressure plate should be in contact with the head, and the tightness should be moderate. The data is read in cm units and is accurate to 0.1.
Weight | The measurement times are before the start of the experiment and the 3rd month after the start
  The weight is measured and obtained by the physician. Place the electronic scale flat on the ground, calibrate the scale reading, instruct the examinee to empty their bowels and bladder, wear light clothing and stand barefoot naturally in the center of the electronic scale pedal, keep the body stable, record the data, the unit is kg, and the value is accurate to 0.1.
Uterine volume | The measurement times are before the start of the experiment and the 3rd month after the start
  Uterine volume obtained through ultrasound measurement; The size and shape of the organs are measured by a professional ultrasound physician from our hospital. The volume is calculated using the formula: V=(π /6)lengthanteroposterior diameter*transverse diameter, with the unit being cubic centimeters (cm³).
Waist-Hip Ratio | The measurement times are before the start of the experiment and the 3rd month after the start
  Use a flexible, non-elastic anthropometric tape (mm-scale) and have the subject stand upright (feet shoulder-width apart, arms relaxed, abdomen relaxed) in lightweight, form-fitting clothing.
  For waist circumference: Mark the midpoint between the costal arch's inferior margin and iliac crest's superior border (umbilicus as alternative if unclear). Wrap the tape horizontally here-level, skin-adherent, no subcutaneous compression. Record to 0.1 cm at end of normal expiration; average 2-3 readings.
  For hip circumference: Locate the gluteal region's widest transverse diameter (confirmed posteriorly/laterally). Wrap tape horizontally here (level, flat). Record to 0.1 cm; average 2-3 readings.
  Compute WHR as mean waist ÷ mean hip (decimal, e.g., 85.2 cm ÷ 102.5 cm ≈ 0.83). Trained personnel must conduct measurements to reduce inter-observer variation.
ovarian volume | The measurement times are before the start of the experiment and the 3rd month after the start
  Ovarian volume obtained through ultrasound measurement The size and shape of the organs are measured by a professional ultrasound physician from our hospital. The volume is calculated using the formula: V=(π /6)lengthanteroposterior diameter*transverse diameter, with the unit being cubic centimeters (cm³).
follicle diameter | The measurement times are before the start of the experiment and the 3rd month after the start
  Follicle diameter obtained through ultrasound measurement The size and shape of the organs are measured by a professional ultrasound physician from our hospital.
Serum levels of various steroid hormones | The measurement times are before the start of the experiment and the 3rd month after the start
  Serum metabolomics sequencing:Liquid Chromatography-Mass Spectrometry (LC-MS) technology for non-targeted metabolomics detection of small-molecule metabolites in serum, and simultaneously using a targeted steroid hormone panel for profiling.
Fecal sample gut microbiota | The measurement times are before the start of the experiment and the 3rd month after the start
  Analysis of gut microbiota detection: detection of gut microbiota in fecal samples (16sRNA, gut microbiome metagenomics, metabolomics).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided